CLINICAL TRIAL: NCT01989650
Title: The Effect of Taking Break During Colonoscopy Session on Adenoma Detection, a Prospective, Randomized Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Aric Josun Hui, Dr., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Break
Record Dates: First submitted 2013-11-07; First posted 2013-11-21 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Colonic Adenoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Break (Active Comparator): A break of 15 minute will be provided after 3rd colonoscopy in a session of 6 colonoscopies in total
  Interventions: Other: Break; Other: No break
- No break (No Intervention): No break will be provided

INTERVENTIONS:
Other: Break — A break of 15 minute will be provided after 3rd colonoscopy in a session of 6 colonoscopies in total
  Arms: Break
Other: No break — No break will be provided
  Arms: Break

SUMMARY:
Recent research has suggested that endoscopist fatigue may significantly affect the polyp detection rate. There have been no studies on interventions that may reduce endoscopist fatigue and therefore improve colonoscopy performance.

We want to determine whether a break in the middle of colonoscopy session would maintain a more stable adenoma detection rate

DETAILED DESCRIPTION:
In recent years, there has been a dramatic increase in the volume of endoscopic procedures performed in most endoscopy centers. With the growing awareness of colorectal cancer screening, there is increasing demand for colonoscopy which has increased the workload of endoscopists in every healthcare system. There are studies showing that physician fatigue impairs quality of care and performance in other medical specialties such as anesthesia and surgery. Colonoscopy by nature is repetitive and frequently prolonged which can promote distractibility and fatigability. Studies from western countries have showed that afternoon colonoscopies are associated with lower adenoma detection rate (ADR) compared with the morning colonoscopies and physician fatigue has been hypothesized as a potential contributor. Previous studies also showed that the polyp detection rate decreases hour-by-hour throughout the day and the colonoscopy completion rate appears to decline with successive procedures due to endoscopist fatigue. The most recent study using the queue position as a surrogate marker for endoscopist fatigue had showed that both the later colonoscopy start time and increasing number of preceding endoscopic procedures are associated with decreasing polyp detection rate. It is not surprising that endoscopist fatigue may contribute to a significant decline in the effectiveness of colonoscopy and yet it is probably not realistic to reduce the number of colonoscopy procedures per session given the heavy clinical demand. There have been no studies on any intervention that may improve the performance of colonoscopy. It would be reasonable to postulate that taking a break half way through the colonoscopy session may alleviate endoscopist fatigue and hence improve the polyp detection rate. This study aims to evaluate the effect of introducing a break in the middle of a colonoscopy session on the quality of colonoscopy performance.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent colonoscopies in the afternoon session at the endoscopy unit in AHNH were eligible for inclusion in this study.

Exclusion Criteria:

* Emergency inpatient colonoscopy
* Patient with history of colorectal cancer , FAP or IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1379 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 2 years

SECONDARY OUTCOMES:
Colonoscopy insertion time | 2 years
Cecal intubation rate | 2 years
Patient satisfaction score | 2 years
  A questionnaire will be used to asses patient's satisfaction level
Complication rate | 2 years
Withdrawal time | 2 years
Patient pain score | 2 years
  A questionnaire will be used to asses patient's level of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hong Kong